CLINICAL TRIAL: NCT03106103
Title: Incidence of Symptomatic and Asymptomatic Bacteriuria After Urodynamic Study With or Without Antibiotic Prophylaxis in Women With Urinary Incontinence
Brief Title: Incidence of Symptomatic and Asymptomatic Bacteriuria After Urodynamic Study in Women
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Elizabeth Yukie Hirakauva, doctor, Federal University of São Paulo
Other Study IDs: EYH-2014
Record Dates: First submitted 2014-06-10; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Female Stress Incontinence
Keywords: urodynamics; cystitis; prophylactic antibiotics; bacteriuria
MeSH Terms: conditions — Cystitis; Bacteriuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women with urinary incontinence: The patients were randomized in four groups: Group A received 500mg of levofloxacin, group B received placebo, group C received 80mg trimethoprim and 400mg sulfamethoxazole (SMZ-TMP) and group D received 100mg of nitrofurantoin.

SUMMARY:
Urodynamic Study (UDS) represents a series of agreed-upon clinical tests and is used to evaluate the functional status of the lower urinary tract, providing a pathophysiological basis for urinary symptoms. Urodynamic Study involves catheterization of the lower urinary tract. The prevalence of urinary tract infection after UDS ranges from 1,5% to 30 %.

Studies of prophylactic antibiotics for UDSs have offered data of contradictory and limited predictive values. Some investigators concluded that prophylactic antibiotics were valuable and others have not.

The objective of this study is to evaluate the efficacy of antibiotic prophylaxis before UDS in women, using different antibiotic regimens.

DETAILED DESCRIPTION:
This study is randomized, double blind study was carried out in the Department of Gynecology at Sao Paulo Federal University from January 2009 to December 2012.

The patients were randomized in four groups: Group A received 500mg of levofloxacin, group B received placebo, group C received 80mg trimethoprim and 400mg sulfamethoxazole (SMZ-TMP) and group D received 100mg of nitrofurantoin. The tablets were administered 30 minutes before de UDS.

All patients were instructed to collect midstream urine sample to the microbiology laboratory 14 days after the UDS. Significant bacteriuria was considered when >1.000.000 organisms/mL of a single species was isolated.

All data were entered into Statistical Package for Social Sciences (SPSS) 16.0 for statistical analysis and graphic representation. Likelihood -ratio test and Fisher's exact test were used to compare the prevalence of significant bacteriuria after UDS in the different groups and Student's t-test and ANOVA test were used to compare continuous variables. To compare the groups regarding the BMI variable and parity, the model analysis of variance (ANOVA) was used, or if necessary, the nonparametric Kruskal-Wallis test and to compare the groups in relation to menopause variable, we used the Chi-square test. A significance level of 0.05 was established for statistical analysis.

ELIGIBILITY:
* Inclusion Criteria: Women with 20 to 85 years old, clinical diagnosis of urinary incontinence with indication for urodynamic study, absence of genital prolapse or prolapse peak effort that does not exceed the hymen, absence of urinary tract infection
* Exclusion Criteria: Patients with diabetes mellitus, history of recurrence urinary tract infection, with genital prolapse that exceed de hymen, pregnant, kidney stone, allergy to antibiotics, use of urethral catheters delay

Ages: 18 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with urinary dysfunction
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic and asymptomatic bacteriuria after urodynamic study in women with urinary incontinence | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hirakauva, Doctor, Principal Investigator — Federal University of São Paulo